CLINICAL TRIAL: NCT04172948
Title: The Utility of Virtual Reality in the Management of Pediatric Functional Constipation With Pelvic Floor Dysfunction.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Lucile Packard Children's Hospital (Other)
Responsible Party: Principal Investigator, Ann Ming Yeh, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52684
Record Dates: First submitted 2019-11-13; First posted 2019-11-21 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Functional Constipation; Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Care Provider
Masking Description: Care provider will be blinded to the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual reality arm (Experimental): This arm will receive diaphragmatic breathing teaching by a medical professional and virtual reality module that teaches diaphragmatic breathing. This arm will be sent home with the virtual reality equipment and practice this breathing technique through the virtual reality module for 8 weeks.
  Interventions: Device: Oculus go headset/virtual reality headset; Behavioral: Diaphragmatic breathing
- Control (Placebo Comparator): This arm will receive diaphragmatic breathing teaching by a medical professional only. They will practice this breathing technique with a paper handout of diaphragmatic breathing technique instructions for 8 weeks.
  Interventions: Behavioral: Diaphragmatic breathing

INTERVENTIONS:
Device: Oculus go headset/virtual reality headset — 10 minute virtual reality tutorial on diaphragmatic breathing, a game in practicing diaphragmatic breathing, and two scenarios in which the patient can also practice diaphragmatic breathing.
  Arms: Virtual reality arm
Behavioral: Diaphragmatic breathing — 10 minute tutorial on diaphragmatic breathing by a medical professional.

SUMMARY:
1. To determine if the adjunctive use of a Virtual Reality (VR) module on diaphragmatic breathing (DB) can improve the quality of life (QOL) and symptoms of children with functional constipation (FC) with pelvic floor dysfunction (PFD) who are receiving standard of care treatment.
2. To assess if a VR module on DB can decrease healthcare utilization for children with FC with PFD.

DETAILED DESCRIPTION:
The investigators will assess if the use a Virtual Reality (VR) module on diaphragmatic breathing (DB) can improve quality of life, constipation symptoms, and decrease healthcare utilization for children with functional constipation (FC) with pelvic floor dysfunction (PFD). FC is a common pediatric condition with a high prevalence and $4.25 billion yearly in healthcare expenditures. FC is often complicated with PFD as seen through stool withholding behaviors. Children with FC with PFD are referred to occupational therapy for biofeedback and DB training as standard of care. Occupational therapy uses to teach children with FC with PFD to relax their abdominal muscles, and subsequently their pelvic floor muscles, facilitating a more complete bowel evacuation. VR is a technology currently employed in rehabilitation services, anesthesiology and surgery. VR can provide a fun, immersive environment with a feedback component for children with FC to learn DB effectively and build a positive association with toileting.

The purpose of this study is to examine if a virtual reality module that teaches children diaphragmatic breathing through an immersive game can improve the quality of life and decrease health care utilization for children with functional constipation and pelvic floor dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Ages 7 to 21 years old
* Meets Rome IV criteria for functional constipation and pelvic floor dysfunction
* Developmentally appropriate to understand verbal instructions

Exclusion Criteria:

* Co-existing medical conditions that include inflammatory bowel disease, Hirschsprung's Disease, cystic fibrosis, tethered cord, anal stenosis, sacral agenesis, spinal cord anomalies, untreated thyroid disease, untreated celiac disease, neurogenic bowel, cerebral palsy, major bowel surgery.
* Non-English speaking

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in baseline in Rome criteria for functional constipation and symptoms of pelvic floor dysfunction. | Baseline, 1 visit between week 2
  This outcome will assess cure of functional constipation and pelvic floor dysfunction.
Change in baseline in Rome criteria for functional constipation and symptoms of pelvic floor dysfunction. | Baseline, week 4
  This outcome will assess cure of functional constipation and pelvic floor dysfunction.
Change in baseline in Rome criteria for functional constipation and symptoms of pelvic floor dysfunction. | Baseline, week 8
  This outcome will assess cure of functional constipation and pelvic floor dysfunction.

SECONDARY OUTCOMES:
Change from baseline in Pediatric Quality of Life (QOL) gastrointestinal (GI) module | Baseline, 1 visit between week 2
  Pediatric Quality of Life Inventory™ Gastrointestinal Symptoms Scales (PedsQL™ Gastrointestinal Symptoms Scales). Scale: 0-4. The total scale score is tallied from the sum of the reversed scores; the higher the score, the higher the health-related quality of life.
Change from baseline in Pediatric Quality of Life (QOL) gastrointestinal (GI) module | Baseline, week 4
  Pediatric Quality of Life Inventory™ Gastrointestinal Symptoms Scales (PedsQL™ Gastrointestinal Symptoms Scales). Scale: 0-4. The total scale score is tallied from the sum of the reversed scores; the higher the score, the higher the health-related quality of life.
Change from baseline in Pediatric Quality of Life (QOL) gastrointestinal (GI) module | Baseline, week 8
  Pediatric Quality of Life Inventory™ Gastrointestinal Symptoms Scales (PedsQL™ Gastrointestinal Symptoms Scales). Scale: 0-4. The total scale score is tallied from the sum of the reversed scores; the higher the score, the higher the health-related quality of life.
Change from baseline in Patient Assessment of Constipation Symptoms (PAC-SYM) constipation questionnaire | Baseline, 1 visit between week 2
  Patient Assessment of Constipation Symptoms (PAC-SYM). The PAC-SYM (12-items) is a survey used to evaluate chronic constipation. Patients rank the symptoms on a 5 point Likert scale, ranging from 0 to 4, 0 being absent and 4 being very severe. For each symptom, score changes of 0.5 points indicate minimal improvement, and changes in 1 point correspond to moderate clinical improvement.
Change from baseline in Patient Assessment of Constipation Symptoms (PAC-SYM) constipation questionnaire | Baseline, week 4
  Patient Assessment of Constipation Symptoms (PAC-SYM). The PAC-SYM (12-items) is a survey used to evaluate chronic constipation. Patients rank the symptoms on a 5 point Likert scale, ranging from 0 to 4, 0 being absent and 4 being very severe. For each symptom, score changes of 0.5 points indicate minimal improvement, and changes in 1 point correspond to moderate clinical improvement.
Change from baseline in Patient Assessment of Constipation Symptoms (PAC-SYM) constipation questionnaire | Baseline, week 8
  Patient Assessment of Constipation Symptoms (PAC-SYM). The PAC-SYM (12-items) is a survey used to evaluate chronic constipation. Patients rank the symptoms on a 5 point Likert scale, ranging from 0 to 4, 0 being absent and 4 being very severe. For each symptom, score changes of 0.5 points indicate minimal improvement, and changes in 1 point correspond to moderate clinical improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Ming Yeh, MD, Principal Investigator — Stanford Hospital/Lucile Packard Children's Hospital; Alice C Huang, MD, Principal Investigator — Stanford Hospital/Lucile Packard Children's Hospital
Locations (1):
- Stanford Hospital/Lucile Packard Children's Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No